CLINICAL TRIAL: NCT05991934
Title: Testing the Impact of Smartphone-based Messaging to Support Young Adult Smoking Cessation
Brief Title: Testing the Impact of Smartphone-based Messaging to Support Young Adult Smoking Cessation - Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00013413-Pilot; IRB00013413 (Other: JHSPH IRB)
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: A pilot micro-randomized trial (within-subject randomization) with 10 young adult smokers will investigate the feasibility of delivering smoking cessation messages based on CBT and mindfulness/ACT for reducing smoking urge 15 minutes after message delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm pilot (Experimental): The micro-randomized trial will determine if CBT and Mindfulness/ACT messages are superior to control messages in reducing the primary outcome momentary smoking urges. Based on participants' training data collected in the initial 14 days of EMA monitoring, intervention messages will be delivered during time-periods and at high-risk locations for smoking. In the intervention phase, participants will be prompted to complete 3 geofence-triggered EMAs per day for a total of 30 days. Each EMA will be followed by an intervention message and the type of message (CBT, Mindfulness/ACT, control) will be randomly selected at each time point (within-subject randomization).
  Interventions: Behavioral: Smartphone-based intervention messages

INTERVENTIONS:
Behavioral: Smartphone-based intervention messages — Intervention messages in the proposed trial will address specific high-risk situations for smoking and smoking urges. Messages will focus on two key situational triggers for message matching: 1. Stress (high/low) and 2. Presence of other smokers (yes/no). For each situation, characterized by a combination of these characteristics, several messages were developed. To improve user engagement with the intervention, all messages contain visual content in form of pictures.

SUMMARY:
Clinical practice guidelines for smoking cessation emphasize cognitive behavioral therapy (CBT) to help patients develop coping strategies for urges. Mindfulness or Acceptance and commitment Therapy (ACT) offer a different approach, which teaches smokers psychological flexibility through accepting negative experiences. While there is evidence for the efficacy of both CBT and Mindfulness/ACT smoking cessation interventions, it is unclear if these approaches are efficacious when implemented in real-time and with young adults. The overall goal of this proposal is to evaluate the efficacy of CBT and Mindfulness/ACT messages for young adults targeted at specific high-risk situations for smoking.

DETAILED DESCRIPTION:
To conduct a pilot trial to test CBT and Mindfulness/ACT intervention message efficacy for reducing momentary smoking urges (N=10). To inform just-in-time interventions, it is crucial to test if CBT and Mindfulness/ACT based messages can reduce momentary smoking urges. The investigators will conduct a micro-randomized trial (repeated within-subject randomizations of messages) to accomplish this. In line with the investigators' existing protocol, participants first collect Ecological Momentary Assessment (EMA) data for 14 days, allowing the investigators to determine high-risk situations for smoking. In the following intervention phase, participants receive tailored messages triggered by geofencing of participants' high-risk locations for a total of 30 days. Tailoring is based on established predictors of smoking relapse (stress and presence of other smokers). The micro-randomized trial tests the efficacy of CBT versus Mindfulness/ACT versus control messages for reducing smoking urge 15 minutes post message delivery. Secondary outcomes include smoking or other tobacco use (including e-cigarettes), affect, and stress. After 45 days, follow up interviews with participants will be conducted to collect information on their study experience.

ELIGIBILITY:
Inclusion Criteria:

1. live in the U.S.
2. read English;
3. are between 18 and 30 years of age;
4. own an iPhone or Android smartphone;
5. have smoked ≥100 cigarettes and currently smoke at least 1 cigarette per day on 3 or more days of the week;
6. are planning to quit smoking within the next 30 days.

Exclusion Criteria:

* live internationally
* don't read English
* younger than 18, older than 30
* don't own a iPhone or Android smartphone
* have smoked less than 100 cigarettes
* not planning to quit smoking in the next 30 days

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Thrul, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Any individual requests for data will be honored on a case-by-case basis as deemed appropriate to the research protocol.

REFERENCES:
- [Derived] Thrul J, Devkota J, Hamoud J, Waring JJC, Luken A, Han JJ, Naughton F, Zipunnikov V, Mendelson T, Latkin C, Moran M, Epstein D, Desjardins MR. Micro-randomized pilot trial of an app-based smoking urge reduction intervention for young adults. Mhealth. 2025 Oct 29;11:59. doi: 10.21037/mhealth-25-17. eCollection 2025. PMID 41211017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through Facebook, Instagram, Reddit, and X advertisements that linked to a Qualtrics screening survey. All participants who met eligibility criteria had to provide online consent prior to study involvement. After consenting to participate but before being enrolled into the study, participants were required to send study staff a picture of a valid identification (e.g., driver's license) that had their name, picture, and birthdate to validate their age and identity.
Period: Overall Study
Arm/Group | Single Arm Pilot
Started | 12
Completed | 8
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Pilot
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Smoking Urge as Assessed by Survey Item
Description: The primary outcome is change in participants' rating of smoking urge from pre- to post-message surveys. Urge is assessed by a single item on a 5-point scale, ranging from 1 (very low) to 5 (very high) in pre and post surveys. Pre-message surveys are completed immediately before message delivery and post-message surveys are prompted 15 minutes after intervention message delivery. . Data presented here are Mean and Standard Deviation of smoking urge before (pre-message EMA) and after (follow-up EMA) a message was delivered for the different message conditions (Control, Cognitive behavioral therapy (CBT), Mindfulness or Acceptance and commitment Therapy (ACT)). Messages were randomized within subjects.
Time Frame: Baseline, 15 minutes after message delivery
Population: A total of 4 participants removed after the initial assessment phase who did not provide required data to construct geo-fences of high-risk situations for smoking that were required for the intervention phase and thus did not advance to the intervention phase and did not receive intervention messages.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Message exposures
Arm/Group | Single Arm Pilot
Number analyzed (Participants) | 8
Number analyzed (Message exposures) | 291
units on a scale
  Control: Pre-message EMA, smoking urge | 2.59 (1.30)
  Control: Follow-up EMA, smoking urge | 2.39 (1.27)
  CBT: Pre-message EMA, smoking urge | 2.53 (1.50)
  CBT: Follow-up EMA, smoking urge | 2.16 (1.35)
  ACT: Pre-message EMA, smoking urge | 2.76 (1.34)
  ACT: Follow-up EMA, smoking urge | 2.40 (1.30)

2. Primary Outcome: Change in Number of Cigarettes Smoked Per Day in Past Week as Assessed by a Single Item
Description: The primary outcome will be change in self-reported number of cigarettes smoked per day in the past week from baseline to 45-days.
Time Frame: Baseline, 45-day follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Arm/Group | Single Arm Pilot
Number analyzed (Participants) | 8
Cigarettes per day
  Baseline | 7.1 (5.8)
  45-day follow-up | 3.2 (2.2)

ADVERSE EVENTS:
Time Frame: Up to 45 days
Arm/Group | Single Arm Pilot
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT05991934/Prot_SAP_000.pdf